CLINICAL TRIAL: NCT03220581
Title: A Psychotherapy Development Study for a New Addictive Disorder
Brief Title: A Psychotherapy Development Study for Internet Gaming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kristyn Zajac, Assistant Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-028-2; R21DA042900 (NIH)
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Referral and Consultation; Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Referral for care (Active Comparator): Referral for mental health issues and family support services
  Interventions: Behavioral: Referral for care
- Behavioral therapy (Experimental): 8-week behavioral intervention designed to assist with better monitoring and regulating the child's game playing behaviors
  Interventions: Behavioral: Referral for care; Behavioral: Behavioral therapy

INTERVENTIONS:
Behavioral: Referral for care — referral for addictions support
Behavioral: Behavioral therapy — therapy focused on monitoring gaming behavior and replacing it with other activities and communication skills
  Arms: Behavioral therapy

SUMMARY:
The fifth edition of the Diagnostic and Statistical Manual for Mental Disorders (DSM-5) introduces Internet Gaming disorder (IGD) as a Substance-Related and Addictive Disorder in Section 3, Conditions for Further Study. Although research is in the nascent stages, existing studies demonstrate that IGD is associated with psychosocial distress including suicidality, and adverse vocational and educational outcomes in youth. Internet gaming disorder also shares substantial overlap with substance use, and it primarily affects adolescents, who rarely seek treatment on their own. Parents more often express concerns about their child's game playing behaviors, and data suggest that parents can have strong influences on it. This psychotherapy development study will evaluate feasibility, acceptability, and effect sizes of a behavioral intervention designed to help parents reduce gaming problems in their children. Sixty concerned parents and their children will complete parental and self-report inventories and structured diagnostic interviews regarding the child's gaming behaviors, substance use and psychosocial functioning. Participants will be randomized to either a control condition consisting of referral for mental health issues and family support services or to the same plus a 6-week family-based behavioral intervention designed to assist with better monitoring and regulating the child's game playing behaviors and encouraging and rewarding alternatives to game playing. Gaming and other problems will be assessed pre-treatment, mid-treatment, at the end of treatment, and at a 4-month follow-up. This study is unique in evaluating initial psychometric properties of a parental version of a measure that uses the DSM-5 criteria for IGD in a clinical sample, and it will also assess associations of IGD with substance use, psychological symptoms, and family functioning over time. Most importantly, this study will be the first randomized trial of an intervention designed to reduce gambling problems, and results are likely to guide future research and treatment efforts related to this condition.

ELIGIBILITY:
Inclusion Criteria:

* parent/guardian of a 10-19 year old residing in the same household >8 months/year
* reports significant problems with game playing

Exclusion Criteria:

* have a condition that may hinder study participation

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristyn Zajac, PhD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Children were required to participate with a parent; therefore, all children had a parent enrolled in the study. A total of 60 dyads were enrolled in the study. The participant flow table represents the number of children enrolled in the study, as they were the primary target of the intervention.
Period: Overall Study
Arm/Group | Referral for Care | Behavioral Therapy
Started | 28 | 32
Completed | 25 | 25
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Referral for Care | Behavioral Therapy | Total
Number analyzed (Participants) | 28 | 32 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 31 | 58
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.18 (2.29) | 13.84 (2.20) | 13.53 (2.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 27 | 32 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 21 | 27 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 21 | 20 | 41
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 28 | 32 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Completed All 6 Sessions
Description: Completion of sessions is an indicator of treatment acceptability and feasibility
Time Frame: 12 weeks
Population: This outcome is only reported for the Behavioral Therapy group because it is not relevant to the Referral to Care group. The Referral to Care group was not assigned to a structured 6 session intervention; thus, this outcome could not be measured in that group.
Measure: Number; unit: percentage of participants
Groups:
- Behavioral Therapy: 6 session behavioral therapy intervention designed to assist with better monitoring and regulating the child's game playing behaviors
  Referral for care: referral for addictions support
  Behavioral therapy: therapy focused on monitoring gaming behavior and replacing it with other activities and communication skills
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 32
percentage of participants | 40.6

2. Primary Outcome: Number of Days of Gaming in Past Week - Reported by Child
Description: Number of days of game playing in past week is an indicator of severity of the gaming problem.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days/week
Groups:
- Behavioral Therapy: 6 session behavioral intervention designed to assist with better monitoring and regulating the child's game playing behaviors
  Referral for care: referral for addictions support
  Behavioral therapy: therapy focused on monitoring gaming behavior and replacing it with other activities and communication skills
Arm/Group | Referral for Care | Behavioral Therapy
Number analyzed (Participants) | 25 | 25
days/week | 5.04 (1.81) | 3.24 (2.28)
Statistical Analysis 1: Comparison: Referral for Care vs Behavioral Therapy; Test type: Superiority; p = .004, ANCOVA; Baseline number of days of game play in the past week was included as a covariate; F = 9.026

3. Primary Outcome: Number of Days of Gaming in the Past Week - Reported by Parent
Description: Number of days of gaming is an indicator of the severity of the gaming problem.
Time Frame: 12 weeks
Population: The participants included in these analyses were all participants who completed the post-treatment (12 week) assessment. This number differs from the Participant Flow module, which reports the number of participants who completed the final follow-up at 24 weeks.
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Referral for Care | Behavioral Therapy
Number analyzed (Participants) | 26 | 25
days/week | 6.19 (1.58) | 4.04 (3.02)
Statistical Analysis 1: Comparison: Referral for Care vs Behavioral Therapy; Test type: Superiority; p = .007, ANCOVA; Covariate = number of days of gaming in the past week at baseline, reported by the parent; F = 7.922

4. Primary Outcome: Number of Symptoms of Internet Gaming Disorder - Assessed Through a Clinical Interview With Child
Description: Examines whether the treatment group showed greater reductions in symptoms of Internet gaming disorder than the control group. Ratings of Internet gaming disorder symptoms were assessed using a clinical interview with the child, conducted by trained assessors blind to treatment condition.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Symptoms at post-treatment
Arm/Group | Referral for Care | Behavioral Therapy
Number analyzed (Participants) | 25 | 26
Symptoms at post-treatment | 1.28 (1.34) | 0.65 (1.09)
Statistical Analysis 1: Comparison: Referral for Care vs Behavioral Therapy; Test type: Superiority; p = .059, ANCOVA; Controlled for number of symptoms of Internet gaming disorder at baseline - assessed through clinical interview with child; F = 3.73

5. Primary Outcome: Number of Symptoms of Internet Gaming Disorder - Assessed Through a Clinical Interview With Parent
Description: Examines whether the treatment group showed greater reductions in symptoms of Internet gaming disorder than the control group. Ratings of Internet gaming disorder symptoms were assessed using a clinical interview with the parent, conducted by trained assessors blind to treatment condition.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Symptoms at post-treatment
Arm/Group | Referral for Care | Behavioral Therapy
Number analyzed (Participants) | 26 | 25
Symptoms at post-treatment | 2.81 (1.81) | 1.84 (1.65)
Statistical Analysis 1: Comparison: Referral for Care vs Behavioral Therapy; Test type: Superiority; p = .095, ANCOVA; Controlled for baseline number of symptoms of Internet gaming disorder, assessed through clinical interview with the parent; F = 2.91

ADVERSE EVENTS:
Time Frame: From baseline to 24 week follow-up
Arm/Group | Referral for Care | Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/32
Other Adverse Events (participants affected / at risk) | 0/28 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Referral for Care (N=28) | Behavioral Therapy (N=32)
Inpatient Hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
There were no major limitations of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT03220581/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT03220581/ICF_001.pdf